CLINICAL TRIAL: NCT02927301
Title: A Phase II, Open-Label, Multicenter, Single-Arm Study to Investigate the Efficacy and Safety of Atezolizumab as Neoadjuvant and Adjuvant Therapy in Patients With Stage IB, II, IIIA, or Selected IIIB Resectable and Untreated Non-Small Cell Lung Cancer
Brief Title: A Study of Atezolizumab as Neoadjuvant and Adjuvant Therapy in Resectable Non-Small Cell Lung Cancer (NSCLC) - Lung Cancer Mutation Consortium (LCMC3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML39236
Record Dates: First submitted 2016-10-05; First posted 2016-10-07 (Estimated); Results first posted 2021-05-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (Experimental): Participants received two cycles of atezolizumab as neoadjuvant therapy prior to surgery. Participants who demonstrated clinical benefit were eligible to receive up to 12 months of atezolizumab.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody — Atezolizumab was given as 1200 milligrams (mg) via intravenous (IV) infusion on Day 1 of each 21-day cycle.
  Other Names: RO5541267, MPDL3280A

SUMMARY:
This study was designed to evaluate the safety and efficacy of neoadjuvant and adjuvant atezolizumab in participants with resectable Non-Small Cell Lung Cancer (NSCLC). Neoadjuvant therapy consisted of two 21-day cycles with atezolizumab. Following surgery, adjuvant therapy consisted of up to 12 months of atezolizumab in participants who demonstrate clinical benefit with neoadjuvant therapy. All participants who undergo surgery entered a surveillance period, which consisted of standardized blood sample collection and Chest CT Scans, for up to 2 years. All participants were monitored for disease recurrence and survival for up to 3 years after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented Stage IB, II, IIIA, or selected IIIB, including T3N2 or T4 (by size criteria, not by mediastinal invasion) NSCLC
* Adequate pulmonary and cardiac function
* Available biopsy of primary tumor with adequate samples
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* NSCLC that is clinically T4 by virtue of mediastinal organ invasion or Stage IIIB by virtue of N3 disease
* Any prior therapy for lung cancer within 3 years.
* Prior treatment with anti-PD-1 or PD-L1 therapies
* History or risk of autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- United States (19):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCLA Cancer Center, Santa Monica, California
  - University Of Colorado, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University; Winship Cancer Institute, Atlanta, Georgia
  - Dana Farber Cancer Institute; Brigham and Womens Hospital, Boston, Massachusetts
  - Mass General/North Shore Cancer, Danvers, Massachusetts
  - Karmanos Cancer Inst; Hematology/Oncology, Detroit, Michigan
  - Washington University; Wash Uni. Sch. Of Med, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering - Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center - Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center at Westchester, Harrison, New York
  - New York University Medical Center, New York, New York
  - Memorial Sloan Kettering - Basking Ridge, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Derived] Chaft JE, Oezkan F, Kris MG, Bunn PA, Wistuba II, Kwiatkowski DJ, Owen DH, Tang Y, Johnson BE, Lee JM, Lozanski G, Pietrzak M, Seweryn M, Byun WY, Schulze K, Nicholas A, Johnson A, Grindheim J, Hilz S, Shames DS, Rivard C, Toloza E, Haura EB, McNamee CJ, Patterson GA, Waqar SN, Rusch VW, Carbone DP; LCMC study investigators. Neoadjuvant atezolizumab for resectable non-small cell lung cancer: an open-label, single-arm phase II trial. Nat Med. 2022 Oct;28(10):2155-2161. doi: 10.1038/s41591-022-01962-5. Epub 2022 Sep 12. PMID 36097216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 181 participants diagnosed with Stage IB, II, IIIA, or selected IIIB resectable and untreated non-small-cell lung cancer (NSCLC) took part in the study in the United States from 20 Apr 2017 to 05 Sep 2023.
Groups:
- Atezolizumab: Participants received atezolizumab, 1200 milligram (mg) as intravenous (IV) infusion, once every 21 days (Q21D) for a maximum of 2 cycles (1 cycle=21 days) as neo-adjuvant therapy. Participants who demonstrated clinical benefit from neo-adjuvant therapy and subsequently underwent surgery then received adjuvant treatment with atezolizumab, 1200 mg, as IV infusion, Q21D for a maximum of 12 months.
Period: Overall Study
Arm/Group | Atezolizumab
Started | 181
Participants Who Had Surgery | 159
Completed | 115
Not Completed | 66
Not completed — Death | 39
Not completed — Lost to Follow-up | 8
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 12
Not completed — Study Ended By Sponsor While in Survival Follow-Up | 5

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who have received any dose of study drug.
Groups:
- Atezolizumab: Participants received atezolizumab, 1200 mg as IV infusion, Q21D for a maximum of 2 cycles (1 cycle=21 days) as neo-adjuvant therapy. Participants who demonstrated clinical benefit from neo-adjuvant therapy and subsequently underwent surgery then received adjuvant treatment with atezolizumab, 1200 mg, as IV infusion, Q21D for a maximum of 12 months.
Arm/Group | Atezolizumab
Number analyzed (Participants) | 181
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.1 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 159
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 145
  More than one race | 0
  Unknown or Not Reported | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Major Pathologic Response (MPR)
Description: Major pathologic response was defined as ≤10% of viable tumor cells as scored by a pathologist, based on surgical resection as defined by prior studies. Percentages have been rounded off to the nearest decimal point.
Time Frame: After surgery (approximately 10 weeks)
Population: The Primary Efficacy Population (PEP) included NSCLC participants who had received surgery after neoadjuvant treatment with atezolizumab, received at least one dose of the study drug, and who did not have Epidermal Growth Factor Receptor (EGFR) or Anaplastic Lymphoma Kinase (ALK) mutant tumors. The overall number analyzed was the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 143
percentage of participants | 20.3
Statistical Analysis 1: Comparison: Atezolizumab; Test type: Superiority; p < .0001, binomial test; Other/Percentage = 20.3, 95% CI 1-sided [lower limit 14.900]

2. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) for PD-L1-Positive Versus PD-L1-Negative Participants
Description: ORR was defined as percentage of participants with complete response (CR) or partial response (PR) as determined by the investigator using RECIST v.1.1, assessed in the programmed death ligand 1 (PD-L1) positive (participants with combined tumor cell (TC)/ immune cell (IC) score categorized as TC1/2/3 or IC1/2/3) and PD-L1 negative (participants with TC/IC score was categorized as TC0 and IC0) groups. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Percentages have been rounded off to the nearest decimal point.
Time Frame: Pre-surgery (Day 36 +/- 3 days), after 2 doses of neoadjuvant treatment with atezolizumab
Population: The overall number analyzed included participants in the PEP with non-missing ORR data and PD-L1 status. The PEP included participants with NSCLC who had received surgery after neoadjuvant treatment with atezolizumab, received at least one dose of the study drug, and who did not have EGFR or ALK mutant tumors. The number analyzed per row was the number of participants with data available for analysis in each PD-L1 group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 112
percentage of participants
  PD-L1 Positive Group: number analyzed (Participants) | 60
  PD-L1 Positive Group | 13.3 [5.9 to 24.6]
  PD-L1 Negative Group: number analyzed (Participants) | 52
  PD-L1 Negative Group | 1.9 [0.1 to 10.3]
Statistical Analysis 1: Comparison: Atezolizumab; Test type: Superiority; p = 0.0358, Fisher Exact; Risk Difference (RD) = 11.410, 80% CI 1-sided [lower limit 5.279]

3. Secondary Outcome: Percentage of Participants With Major Pathologic Response for PD-L1-Positive Versus PD-L1-Negative Participants
Description: Major pathologic response (MPR) was defined as ≤10% of viable tumor cells, as scored by a pathologist, based on surgical resection as defined by prior studies. MPR was assessed based on participants tumor cell (TC) and immune cell (IC) score. The participants were considered as PD-L1- positive if their combined TC/IC score was categorized as TC1/2/3 or IC1/2/3 and the participants were considered PD-L1 negative if TC/IC score was categorized as TC0 and IC0. Percentages have been rounded off to the nearest decimal point.
Time Frame: After surgery (approximately 10 weeks)
Population: The overall number analyzed included participants in the PEP with non-missing MPR data and PD-L1 status. PEP included participants with NSCLC who had received surgery after neoadjuvant treatment with atezolizumab, received at least one dose of the study drug, and who did not have EGFR or ALK mutant tumors. The number analyzed per row was the number of participants with data available for analysis in each PD-L1 group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 109
percentage of participants
  PD-L1 Positive Group: number analyzed (Participants) | 57
  PD-L1 Positive Group | 29.8 [18.4 to 43.4]
  PD-L1 Negative Group: number analyzed (Participants) | 52
  PD-L1 Negative Group | 13.5 [5.6 to 25.8]
Statistical Analysis 1: Comparison: Atezolizumab; Test type: Superiority; p = 0.0395, Chi-squared; Risk Difference (RD) = 16.363, 80% CI 1-sided [lower limit 6.509]

4. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: An adverse event (AE) was defined as any untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product. AEs were reported based on the National Cancer Institute Common Terminology Criteria for AEs, version 4.0 (NCI-CTCAE, v4.0).
Time Frame: From first study dose of atezolizumab until 90 days after the last study dose of atezolizumab (up to 18 months)
Population: Safety population included all enrolled NSCLC participants who have received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 181
Participants | 177

5. Secondary Outcome: Percentage of Participants With Major Pathologic Response (MPR) by Mutation Load
Description: MPR was defined as ≤10% of viable tumor cells in the surgical resection as scored by a pathologist. Whole-exome sequencing (WES) was run, and the consequences of each mutation were determined using Ensembl Variant Effect Predictor (VEP). Mutation load (i.e. tumor mutation burden (TMB)) was defined as the number of variants altering protein sequence as outlined by VEP divided by 34 Megabase (MB) of assay target region. The final value was reported as number of mutations per megabase (mut/MB). It was divided into three groups: TMB <10 mut/MB; TMB ≥ 10 mut/MB to <16 mut/MB; and TMB ≥16 mut/MB. Percentages have been rounded off to the nearest decimal point.
Time Frame: Up to 13 weeks
Population: The overall number analyzed included participants in the PEP with non-missing MPR and TMB data. The PEP included participants with NSCLC who had received surgery after neoadjuvant treatment with atezolizumab, received at least one dose of the study drug, and who did not have EGFR or ALK mutant tumors. The number analyzed per row is the number of participants with data available for analysis in each TMB subgroup.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 86
percentage of participants
  TMB <10 mut/MB: number analyzed (Participants) | 60
  TMB <10 mut/MB | 16.7 [8.3 to 28.5]
  TMB ≥10 mut/MB to <16 mut/MB: number analyzed (Participants) | 11
  TMB ≥10 mut/MB to <16 mut/MB | 9.1 [0.2 to 41.3]
  TMB ≥16 mut/MB: number analyzed (Participants) | 15
  TMB ≥16 mut/MB | 33.3 [11.8 to 61.6]

6. Secondary Outcome: Percentage of Participants With Major Pathologic Response (MPR) by Neoantigen Score
Description: MPR was defined as ≤10% of viable tumor cells in the surgical resection as scored by a pathologist. MPR was analysed by neoantigen score, which was assessed based on the number of highly immunogenic, expressed neoantigens detected at baseline. Median splits were applied for analyses of MPR. Neoantigen scores >/= 73 (i.e. >/= 73 highly immunogenic, expressed neoantigens detected at baseline) were considered as high scores, and scores <73 (i.e. <73 highly immunogenic, expressed neoantigens detected at baseline) were considered as low neoantigen scores. Percentages have been rounded off to the nearest decimal point.
Time Frame: Up to 13 weeks
Population: The overall number analyzed included participants in the PEP with non-missing MPR and neoantigen score data. The PEP included those with NSCLC who had received surgery after neoadjuvant treatment with atezolizumab, received at least one dose of the study drug, and who did not have EGFR or ALK mutant tumors. The number analyzed per row is the number of participants with data available for analysis in each neoantigen score subgroup.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 62
percentage of participants
  Low score: number analyzed (Participants) | 31
  Low score | 19.4 [7.5 to 37.5]
  High score: number analyzed (Participants) | 31
  High score | 25.8 [11.9 to 44.6]

7. Secondary Outcome: Percentage of Participants With Major Pathologic Response (MPR) by Gene Expression Signatures: Gene Set Variation Analysis (GSVA)
Description: MPR was defined as ≤10% of viable tumor cells in the surgical resection as scored by a pathologist. MPR was analysed by gene set variation analysis (GSVA) scores. Bulk ribonucleic acid (RNA) from baseline tumor samples were assessed using GSVA for a T effector cell (Teff) signature comprising the following genes: cluster of differentiation 8A (CD8A), eomesodermin (EOMES), granzyme A (GZMA), T-box transcription factor 21 (TBX21), interferon-gamma (IFNG), granzyme B (GZMB), C-X-C motif chemokine ligand 9 (CXCL9), and C-X-C motif chemokine ligand 10 (CXCL10). Tertile splits were applied to GSVA scores, categorized as lower, middle, and upper scores, which indicated the relative levels of gene set expression in the baseline tumor samples. Percentages have been rounded off to the nearest decimal point.
Time Frame: Up to 13 weeks
Population: The overall number analysed included participants in the PEP with non-missing MPR and GSVA score data. The PEP included participants with NSCLC who had received surgery after neoadjuvant treatment with atezolizumab, received at least one dose of the study drug, and who did not have EGFR or ALK mutant tumors. The number analyzed per row was the number of participants with data available for analysis in each GSVA score subgroup.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 52
percentage of participants
  Lower score: number analyzed (Participants) | 17
  Lower score | 17.6 [3.8 to 43.4]
  Middle score: number analyzed (Participants) | 17
  Middle score | 35.3 [14.2 to 61.7]
  Upper score: number analyzed (Participants) | 18
  Upper score | 33.3 [13.3 to 59.0]

8. Secondary Outcome: Percentage of Participants With Major Pathologic Response (MPR) by Gene Expression Signatures: xCell Immune Score
Description: MPR was defined as ≤10% of viable tumor cells in the surgical resection as scored by a pathologist. MPR was analysed by gene expression signatures. Bulk RNA from baseline tumor samples were assessed using xCell immune score. Tertile splits were applied to xCell immune scores, categorized as lower, middle, and upper scores, which indicated the relative levels of immune cell gene expression in the baseline tumor samples. Percentages have been rounded off to the nearest decimal point.
Time Frame: Up to 13 weeks
Population: The overall number analyzed included participants in the PEP with non-missing MPR and xCell immune score data. The PEP included participants with NSCLC who had received surgery after neoadjuvant treatment with atezolizumab, received at least one dose of the study drug, and who did not have EGFR or ALK mutant tumors. The number analyzed per row was the number of participants with data available for analysis in each xCell immune score subgroup.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 52
percentage of participants
  Lower score: number analyzed (Participants) | 17
  Lower score | 29.4 [10.3 to 56.0]
  Middle score: number analyzed (Participants) | 17
  Middle score | 23.5 [6.8 to 49.9]
  Upper score: number analyzed (Participants) | 18
  Upper score | 33.3 [13.3 to 59.0]

ADVERSE EVENTS:
Time Frame: Adverse events: From first study dose of atezolizumab until 90 days after the last study dose of atezolizumab (up to 18 months); All-cause mortality: From first dose of study treatment until end of follow-up (up to 59 months)
Description: Safety population included all enrolled NSCLC participants who have received any dose of study drug.
Arm/Group | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 39/181
Serious Adverse Events (participants affected / at risk) | 63/181
Other Adverse Events (participants affected / at risk) | 168/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=181)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (4)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Empyema (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 9 (10)
Sepsis (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Sudden death (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Device leakage (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=181)
Anaemia (Blood and lymphatic system disorders) | 19 (19)
Constipation (Gastrointestinal disorders) | 39 (43)
Diarrhoea (Gastrointestinal disorders) | 32 (39)
Nausea (Gastrointestinal disorders) | 40 (49)
Vomiting (Gastrointestinal disorders) | 18 (21)
Upper respiratory tract infection (Infections and infestations) | 11 (12)
Urinary tract infection (Infections and infestations) | 12 (14)
Infusion related reaction (Injury, poisoning and procedural complications) | 16 (17)
Procedural pain (Injury, poisoning and procedural complications) | 54 (55)
Alanine aminotransferase increased (Investigations) | 14 (15)
Aspartate aminotransferase increased (Investigations) | 15 (16)
Weight decreased (Investigations) | 12 (14)
Decreased appetite (Metabolism and nutrition disorders) | 38 (41)
Dehydration (Metabolism and nutrition disorders) | 13 (14)
Hyperkalaemia (Metabolism and nutrition disorders) | 10 (11)
Hyponatraemia (Metabolism and nutrition disorders) | 18 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (45)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (23)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Dizziness (Nervous system disorders) | 21 (22)
Dysgeusia (Nervous system disorders) | 10 (11)
Headache (Nervous system disorders) | 29 (33)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (13)
Anxiety (Psychiatric disorders) | 15 (15)
Insomnia (Psychiatric disorders) | 20 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 36 (40)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 (44)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 11 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 18 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 26 (28)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 (21)
Hypertension (Vascular disorders) | 13 (15)
Hypotension (Vascular disorders) | 12 (12)
Chills (General disorders) | 14 (15)
Fatigue (General disorders) | 79 (93)
Non-cardiac chest pain (General disorders) | 11 (11)
Oedema peripheral (General disorders) | 14 (19)
Pain (General disorders) | 10 (13)
Pyrexia (General disorders) | 25 (26)
Weight increased (Investigations) | 10 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT02927301/Prot_002.pdf
  • Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT02927301/SAP_003.pdf